CLINICAL TRIAL: NCT00215696
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy of BIOBYPASS® (ADGVVEGF121.10NH) Delivered by NOGA™-GUIDED/MYOSTAR™ Catheter in "No Option" Patients With Class II-IV Stable Angina
Brief Title: A Study to Treat Patients Whose Chronic Angina Symptoms Are Not Relieved by Medication and Have an Area of the Heart That Cannot be Treated by Standard Therapies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GenVec (Industry)
Responsible Party: Paul Fischer, PhD, GenVec
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: GV-002.001
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Moderate to Severe Angina Pectoris

INTERVENTIONS:
Genetic: BioBypass®

SUMMARY:
The primary purpose of this study is to determine whether treatment with an experimental gene therapy (BIOBYPASS®) will reduce angina in study participants by stimulating the growth of new blood vessels. This will be measured by testing whether participants are able to exercise longer without experiencing angina after treatment, as compared to before treatment.

Additionally, this study will collect information about any side effects that might be related to the treatment with the experimental therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years and less than or equal to 80 years;
* Written informed consent obtained prior to any study dictated procedure;
* Moderate to severe angina (CCS Angina Class II-IV) despite optimal medical therapy;
* Treated with optimal unchanged antianginal medical therapy for at least 2 months prior to the first baseline ETT. Optimal medical therapy must include the following medications (unless hemodynamic parameters or intolerance contraindicate their use):

  * Nitroglycerine;
  * Antianginal medications: Long-acting nitrates, calcium-channel blockers, potassium channel opener and beta-blockers (Note: All participants are required to be on at least 2 of the 4 antianginal medications listed above);
  * Platelet aggregation inhibitor (e.g., aspirin, ticlopidine, or clopidogrel)
  * ACE inhibitor
  * Statin (HMG-CoA Reductase Inhibitor)
* The participant must have, within 3 months prior to randomization, documented coronary angiographic evidence of significant 2- or 3- vessel disease, or equivalent disease in one dominant artery, and at least one remaining larger coronary vessel from which new collaterals/vessels could be supplied.
* Any participant who has undergone CABG or PCI within 6 months of entry must have angiography performed within 1 month prior to entry, and at least 4 months after the previous intervention to rule out early restenosis.
* Candidates must not be eligible for any other re-vascularization procedures. The participant and his coronary film must have been discussed with an independent cardiac surgeon and must have been denied for CABG or PTCA. Participants who are marginal or poor candidates for conventional revascularization will be considered eligible if the risks of performing a CABG or PTCA procedure outweigh the potential benefit and/or such a procedure is unlikely to offer a worthwhile clinical benefit. The criteria defining such cases may include, but may not be limited to, the following examples:

  * Diffuse or distal vessel disease
  * Chronic occlusions
  * Unprotected left main stenosis
  * Tortuous or severely angulated vessels
  * Severely calcified vessels
  * Small vessels (< 2.5mm)
* Two baseline bicycle ergometry exercise tolerance tests (ETTs) performed meeting the following criteria:

  * Able to exercise for a minimum duration of 2 minutes and no more than 8 minutes
  * Exercise duration on the two ETTs must be within 15% of each other. (The second test will be used for the baseline value. In the event of excessive variability, a third test may be performed and the participant may be enrolled if exercise duration on the third test is within 15% of either prior test. In this case, the third test will be used as the baseline value.)
  * ETTs must not be discontinued for any reason other than ETT Angina Level 3
  * Note: Participant must NOT be informed of exercise restrictions required for entry.
* Significant reversible myocardial ischemia on a single photon emission computer tomography (SPECT). Judgment will be made by an independent core lab. The size of the reversible defect must be > 10 % of left ventricle.
* Ventricular wall thickness of the treatment zone > 8mm as per baseline echocardiogram.

Exclusion Criteria:

* Pregnant or lactating women. It is required that both men and women use condoms or another barrier method of birth control for at least 8 weeks following administration of BIOBYPASS® and some form of birth control for at least one year;
* Clinically significant anemia (e.g. hematocrit < 36% or hemoglobin < 12 g/dL for men and < 11 g/dL for women), leukopenia (WBC<3,000/µL), leukocytosis (WBC > 12,000), or thrombocytopenia (platelet count < 100,000 billion/l);
* Abnormal prothrombin or partial thromboplastin time or anticoagulant therapy that cannot be withheld for treatment;
* Significant renal dysfunction (serum creatinine > 1.6 mg/dL);
* Hepatic dysfunction (AST/ALT must be within normal limits);
* Hematuria, unless of known, non-malignant etiology (any unexplained hematuria would require the candidate to be excluded);
* Uncontrolled hypertension (systolic blood pressure >200 mmHg or diastolic blood pressure >110 mmHg) or significant hypotension (systolic blood pressure <90 mmHg);
* Conditions other than angina that will limit exercise test (e.g. severe peripheral vascular disease, COPD);
* Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination.

  * Cataract surgery within 6 months of trial;
  * Vascular lesions of the anterior segment of the eye (infection or ulceration of the cornea, rubeotic glaucoma, etc);
  * Vascular lesions of the posterior segment of the eye or proliferative retinopathy in diabetics, macular edema, s/p photocoagulation for macular edema or proliferative retinopathy; nondiabetics with central or branch retinal vascular occlusions, sickle cell retinopathy, ischemic retinopathy due to retinal venous stasis or carotid artery disease);
  * Choroidal new vessels associated with age-related macular degeneration, myopic degeneration, presumed ocular histoplasmosis syndrome, angioid streaks, pseudoxanthoma elasticum, or without ocular disease; and
  * Large elevated choroidal nevi, choroidal vascular tumors (choroidal hemangioma), or melanomas.
* Any acute illness within one week of the start of the study or any other illness considered by the Investigator to significantly interfere with study outcome;
* Clinical evidence of active infection of any type, including adenovirus (evidenced by a screening adenovirus neutralizing antibody titer of > 1:50);
* Immunocompromised status (in the investigator's opinion) or currently receiving immunosuppressive therapy;
* Left ventricular ejection fraction < 25% as measured by LV angiography.
* Congestive heart failure NYHA class III-IV;
* Valvular heart disease requiring surgical intervention or hemodynamically significant aortic valve disease;
* Recent (less than 6 weeks prior to screening) Acute Coronary Syndrome with increase in CK-MB or Troponins/PCI/CABG/Stroke or TIA;
* History of malignancy (except cured non-melanoma skin cancer) or suspicion of current malignancy;
* Known allergy to the diluent used to suspend the virus;
* Other experimental medications within the last four weeks prior to the second baseline ETT;
* Revascularization procedure (percutaneous coronary intervention or coronary artery bypass) within 4 months of Day 1.
* Participants who have previously received VEGF or any other angiogenic agent or gene therapy in the past, or who have participated in other investigational studies within the last year if the endpoints are overlapping.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129
Dates: Start 2005-04

PRIMARY OUTCOMES:
Change from baseline in total exercise duration on exercise tolerance test (ETT, using the bicycle ergometry test protocol) at week 26.

SECONDARY OUTCOMES:
Change of reversible perfusion defect size in SPECT perfusion study at week 26
Total exercise duration at weeks 12 and 52
Time-to-onset of 1mm ST depression on ETT at weeks 12, 26, 52
Peak rate-pressure product and maximal workload (in METS) during ETT at weeks 12, 26, 52
CCS class at weeks 12, 26, 52
Frequency of angina attacks at weeks 12, 26, 52
Nitroglycerine consumption at weeks 12, 26, 52
Results of Seattle angina questionnaire at weeks 12, 26, 52

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jens Kastrup, Principal Investigator — The Heart Center, University hospital Rigshospitalet
Locations (3):
- Denmark (2):
  - Skejby Sygehus, Caridology Laboratory, Århus N
  - Cardiovascular Laboratory 2014, The Heart Center, University hospital Rigshospitalet, Copenhagen
- Cardiac Catheterization Laboratories, Cardiology Department, Rabin Medical Center, Petah, Tikva, Israel